CLINICAL TRIAL: NCT04357067
Title: Comparison of the Clinical Efficacy of the Lingual Brackets and Labial Brackets in the Leveling Phase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, YAZGI AY UNUVAR, PhD, Assistant Professor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DHF-15010
Record Dates: First submitted 2020-04-19; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Irregular Teeth
Keywords: Customized lingual brackets; lingual orthodontics; digital model
MeSH Terms: conditions — Tooth Abnormalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lingual brackets (Experimental): Patients with moderate crowding without extraction treated with Incognito lingual bracket (3M Unitek, Bad Essen, Germany)
  Interventions: Device: Lingual brackets; Device: Labial brackets
- Labial brackets (Experimental): Patients with moderate crowding without extraction treated with labial bracket (3M Unitek, Ca, USA
  Interventions: Device: Lingual brackets; Device: Labial brackets

INTERVENTIONS:
Device: Lingual brackets — A type of bracket that applied lingual surface of teeth.
  Other Names: Customized lingual brackets
Device: Labial brackets — A type of bracket that applied labial surface of teeth.
  Other Names: Conventional labial brackets

SUMMARY:
This aim study aims to compare clinical effectiveness of customized lingual brackets and conventional labial brackets in alignment period in a sample of Class I malocclusion patients treated on a nonextraction basis.

DETAILED DESCRIPTION:
The study included 20 patients who presented with Class I malocclusion and scheduled for orthodontic treatment without tooth extraction. The patients were randomly assigned for treatment with customized lingual brackets or with conventional labial brackets. During the alignment period 0.012 inch (T1) , 0.014 inch(T2), 0.016 inch (T3)NiTi arch wires were performed respectively and the control visits were scheduled by 6-weeks intervals. In all sessions, digital models were obtained by intra-oral scanning device after removal of arch wire, which then analyzed by software. In order to analyze change in T0 (pretreatment), T1, T2 and T3; Little's irregularity index, distance between canine teeth, distance between first premolar teeth, distance between second premolar teeth, distance between first molar teeth and arch length measurements were performed on digital models.

ELIGIBILITY:
Inclusion Criteria:

* Class I malocclusion
* Completed permanent dentition
* Crowding ≥ 6 mm

Exclusion Criteria:

* Tooth loss or extraction except third molars
* Having cross bite
* Having genetic or hormonal disorder
* Using a chronic drug
* Previous orthodontic treatment and prosthetic restoration
* Inappropriate oral hygiene and periodontal diseases

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-01-05 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Irregularity index (mm) | 18 weeks
  Crowding of anterior teeth changes after alignment
Distance between canine teeth (mm) | 18 weeks
  Measurement from right canine to left canine distance
Distance between first premolar teeth (mm) | 18 weeks
  Measurement from right first premolar to left first premolar distance
Distance between second premolar teeth (mm) | 18 weeks
  Measurement from right first premolar to left first premolar distance
Distance between first molar teeth (mm) | 18 weeks
  Measurement from right first molar to left first molar distance

SECONDARY OUTCOMES:
Arch length (mm) | 18 weeks
  Measurement of arch length from mesial side of right first molar to messiah side of left first molar

CONTACTS AND LOCATIONS:
Overall Officials: Yazgı Ay Ünüvar, PhD, Study Director — Aydın Adnan Menderes University Faculty of Dentistry Department of Orthodontics

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khattab TZ, Hajeer MY, Farah H, Al-Sabbagh R. Maxillary dental arch changes following the leveling and alignment stage with lingual and labial orthodontic appliances: a preliminary report of a randomized controlled trial. J Contemp Dent Pract. 2014 Sep 1;15(5):561-6. doi: 10.5005/jp-journals-10024-1579. PMID 25707826
- [Background] Auluck A. Lingual orthodontic treatment: what is the current evidence base? J Orthod. 2013 Sep;40 Suppl 1:S27-33. doi: 10.1179/1465313313Y.0000000073. PMID 24005948
- [Background] Alobeid A, El-Bialy T, Reimann S, Keilig L, Cornelius D, Jager A, Bourauel C. Comparison of the efficacy of tooth alignment among lingual and labial brackets: an in vitro study. Eur J Orthod. 2018 Nov 30;40(6):660-665. doi: 10.1093/ejo/cjy005. PMID 29546390
- [Background] Ziebura T, Hohoff A, Flieger S, Stamm T. Accidental debondings: Buccal vs fully individualized lingual multibracket appliances. Am J Orthod Dentofacial Orthop. 2014 May;145(5):649-54. doi: 10.1016/j.ajodo.2013.12.030. PMID 24785929
- [Background] Sifakakis I, Pandis N, Makou M, Eliades T, Katsaros C, Bourauel C. A comparative assessment of torque generated by lingual and conventional brackets. Eur J Orthod. 2013 Jun;35(3):375-80. doi: 10.1093/ejo/cjs029. Epub 2012 May 9. PMID 22573909
- [Background] Sifakakis I, Pandis N, Makou M, Katsaros C, Eliades T, Bourauel C. A comparative assessment of forces and moments generated by lingual and conventional brackets. Eur J Orthod. 2013 Feb;35(1):82-6. doi: 10.1093/ejo/cjr048. Epub 2011 Apr 4. PMID 21464153
- [Background] Fuck LM, Wiechmann D, Drescher D. Comparison of the initial orthodontic force systems produced by a new lingual bracket system and a straight-wire appliance. J Orofac Orthop. 2005 Sep;66(5):363-76. doi: 10.1007/s00056-005-0442-3. English, German. PMID 16231112